CLINICAL TRIAL: NCT01802151
Title: Evaluation of Bacillus Subtilis R0179 in Capsules on Gastrointestinal Survival, Transit Time, Gastrointestinal Symptoms, and General Wellness in Healthy Young Adults
Brief Title: Evaluation of Bacillus Subtilis R0179 in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Human Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 177-2012
Record Dates: First submitted 2013-02-20; First posted 2013-03-01 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: probiotics; microbiota; survival; gastrointestinal; wellness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (starch, magnesium stearate, citric acid) capsules once daily for 4 weeks.
  Interventions: Dietary Supplement: Placebo
- B. subtilis R0179 (10 billion CFU) (Experimental): B. subtilis R0179 (approximately 10 billion CFU/capsule) once daily for 4 weeks.
  * CFU (Colony Forming Unit)
  Interventions: Dietary Supplement: B. subtilis R0179
- B. subtilis R0179 (1 billion CFU) (Experimental): B. subtilis R0179 (approximately 1 billion CFU/capsule) once daily for 4 weeks.
  Interventions: Dietary Supplement: B. subtilis R0179
- B. subtilis R0179 (0.1 billion CFU) (Experimental): B. subtilis R0179 (approximately 0.1 billion CFU/capsule) once daily for 4 weeks.
  Interventions: Dietary Supplement: B. subtilis R0179

INTERVENTIONS:
Dietary Supplement: B. subtilis R0179 — B. subtilis R0179 for a period of 4 weeks. One capsule per day.
  Arms: B. subtilis R0179 (0.1 billion CFU); B. subtilis R0179 (1 billion CFU); B. subtilis R0179 (10 billion CFU)
Dietary Supplement: Placebo — Placebo (starch, magnesium stearate, citric acid) capsules for a period of 4 weeks. One capsule per day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of three doses of the probiotic B. subtilis (Bacillus subtilis R0179) delivered in capsules on gastrointestinal and general wellness in healthy young adults, survival through the gastrointestinal tract and impact on intestinal microbes.

DETAILED DESCRIPTION:
A 6 week randomized, double blind placebo controlled trial in healthy young adults aged 18 to 50. Participants will be administered an oral dose of B. subtilis or placebo (1 capsule/day) for a period of 4 weeks. Viable counts will be measured from stool samples to assess transit survival, daily questionnaires (DQ) will be administered to assess general wellness, and gastrointestinal (GI) symptoms will be evaluated three times with the Gastrointestinal Symptom Response Scale (GSRS) questionnaire.

ELIGIBILITY:
Inclusion Criteria: Participants

* Are 18-50 years of age
* Are willing and able to complete the Informed Consent Form in English
* Are willing to complete the GPAQ (Global Physical Activity Questionnaire) at baseline and during the last week of the study as well as completing the GSRS (Gastrointestinal Symptom Response Survey) questionnaire at baseline, during treatment and post treatment
* Are currently "moderately active" as determined by the GPAQ (Global Physical Activity Questionnaire)
* Are willing to have height and weight measured and to provide demographic information (age, race, sex)
* Are willing to consume B. subtilis R0179 (approximate doses of 1, 10, or 0.1 billion CFU per day) or placebo for a 28 day period by capsule (1 per day)
* Are willing to complete daily questionnaires regarding general and gastrointestinal wellness for the duration of the study
* Are willing to provide 1 stool at baseline, 1 stool during week 4 of the treatment and 1 stool after 7 days of washout
* Are willing to provide a social security number to receive study payment. Note: the subject can still participate if unwilling to provide social security number, but no financial reimbursement can be provided
* Are willing to have internet access for the duration of the study

Exclusion Criteria: Potential Participants will be excluded if they

* Do not meet the inclusion criteria
* Are currently taking medications for constipation or diarrhea
* Have taken antibiotics within the past four weeks prior to randomization
* Are currently taking probiotics supplements and do not want to discontinue a minimum of two weeks prior to the study
* Known to have or are currently being treated for any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's, ulcerative colitis, etc.), other chronic diseases (diabetes, kidney disease, etc.) or immune-compromising diseases or conditions (HIV, AIDS, autoimmune, hepatitis, cancer, transplant patient etc.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, RD, Principal Investigator — University of Florida; Bobbi Henken-Langkamp, PhD, RD, Principal Investigator — University of Florida; Volker Mai, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Hong HA, Duc le H, Cutting SM. The use of bacterial spore formers as probiotics. FEMS Microbiol Rev. 2005 Sep;29(4):813-35. doi: 10.1016/j.femsre.2004.12.001. Epub 2004 Dec 16. PMID 16102604
- [Background] Oelschlaeger TA. Mechanisms of probiotic actions - A review. Int J Med Microbiol. 2010 Jan;300(1):57-62. doi: 10.1016/j.ijmm.2009.08.005. Epub 2009 Sep 23. PMID 19783474
- [Background] Sanders ME, Morelli L, Tompkins TA. Sporeformers as Human Probiotics: Bacillus, Sporolactobacillus, and Brevibacillus. Compr Rev Food Sci Food Saf. 2003 Jul;2(3):101-110. doi: 10.1111/j.1541-4337.2003.tb00017.x. PMID 33451235
- [Background] Tompkins TA, Hagen KE, Wallace TD, Fillion-Forte V. Safety evaluation of two bacterial strains used in Asian probiotic products. Can J Microbiol. 2008 May;54(5):391-400. doi: 10.1139/w08-022. PMID 18449224
- [Background] Tompkins TA, Xu X, Ahmarani J. A comprehensive review of post-market clinical studies performed in adults with an Asian probiotic formulation. Benef Microbes. 2010 Mar;1(1):93-106. doi: 10.3920/BM2008.1005. PMID 21840798
- [Derived] Hanifi A, Culpepper T, Mai V, Anand A, Ford AL, Ukhanova M, Christman M, Tompkins TA, Dahl WJ. Evaluation of Bacillus subtilis R0179 on gastrointestinal viability and general wellness: a randomised, double-blind, placebo-controlled trial in healthy adults. Benef Microbes. 2015 Mar;6(1):19-27. doi: 10.3920/BM2014.0031. PMID 25062611
- See also: Evaluation of Bacillus subtilis R0179 on gastrointestinal viability and general wellness: a randomised, double-blind, placebo-controlled trial in healthy adults. — http://www.ncbi.nlm.nih.gov/pubmed/25062611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited by flyers and word of mouth on the University of Florida campus. Rolling recruitment (7/02/2012-08/23/2012) occurred until the minimum number of participants (n=80) had been enrolled.
Pre-assignment Details: A one week baseline period was to be completed before participants were randomized to intervention arms. Participants that failed to complete study requirements during this period were withdrawn due to noncompliance.
Groups:
- B. Subtilis R0179 (10 Billion CFU): B. subtilis R0179 (approximately 10 billion CFU/capsule) once daily for 4 weeks.
  B. subtilis R0179: B. subtilis R0179 for a period of 4 weeks. One capsule per day.
Period: Overall Study
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Started | 20 | 21 | 22 | 20
Completed | 20 (Participants were enrolled and randomized in five waves. The final wave's data collection ended 9/20) | 21 (Participants were enrolled and randomized in five waves. The final wave's data collection ended 9/20) | 20 (Participants were enrolled and randomized in five waves. The final wave's data collection ended 9/20) | 20 (Participants were enrolled and randomized in five waves. The final wave's data collection ended 9/20)
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed all study requirements were included in the baseline analysis population. 2 participants in the 1 Billion CFU group were excluded from the baseline analysis because they did not complete all study requirements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU) | Total
Number analyzed (Participants) | 20 | 21 | 20 | 20 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 20 | 20 | 81
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23 [20 to 46] | 23 [20 to 49] | 22 [20 to 31] | 23 [19 to 46] | 23 [19 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 8 | 10 | 42
  Male | 9 | 8 | 12 | 10 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 7 | 2 | 2 | 13
  Black | 4 | 2 | 2 | 2 | 10
  Hispanic | 3 | 2 | 3 | 2 | 10
  White | 9 | 9 | 13 | 14 | 45
  Other | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 20 | 20 | 81
BMI Percentiles [Number; unit: participants]
  <85th % (Healthy Weight) | 10 | 12 | 13 | 9 | 44
  85th-94th % (Overweight) | 6 | 7 | 4 | 9 | 26
  >= 95th % (Obese) | 4 | 2 | 3 | 2 | 11
Activity Level [Mean (Standard Deviation); unit: mins of moderate and intense activity] — Minutes of physical activity were assessed according the Global Physical Activity Questionnaire
  mins of moderate and intense activity | 185.5 (70.9) | 197.3 (84.5) | 168.3 (74.9) | 199.0 (57.9) | 185.9 (72.4)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for GI Distress
Description: Daily Questionnaires consists of 24 symptom items evaluating general wellness. Participants filled out questionnaires nightly for the entire duration of the study (6 weeks). Daily scores were then averaged into weekly scores for each participant. Rating is scored from 0 (no symptoms) to 6 (very severe symptoms).
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (GI Distress) Week 1 | 0.5 (0.8) | 0.3 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Daily Questionnaire (GI Distress) Week 2 | 0.5 (0.1) | 0.4 (0.1) | 0.6 (0.1) | 0.5 (0.1)
  Daily Questionnaire (GI Distress) Week 3 | 0.6 (0.1) | 0.3 (0.1) | 0.6 (0.1) | 0.6 (0.1)
  Daily Questionnaire (GI Distress) Week 4 | 0.6 (0.1) | 0.3 (0.01) | 0.7 (0.1) | 0.7 (0.1)
  Daily Questionnaire (GI Distress) Week 5 | 0.6 (0.1) | 0.3 (0.1) | 0.7 (0.1) | 0.5 (0.1)
  Daily Questionnaire (GI Distress) Week 6 | 0.5 (0.1) | 0.3 (0.1) | 0.6 (0.1) | 0.4 (0.1)

2. Secondary Outcome: Evaluation of the Survival of B. Subtilis R0179 and Analyzing the Microbial Diversity in Stool Samples by Participants (Microbiota Study)
Description: Viability of B. subtilis R0179, recovered from stool samples, was assessed using one way ANOVA followed subsequently by Tukey-Kramer HSD when significance was reached (p<0.05). Data was normalized when appropriate. Data analyzed was log (CFU/g).
Time Frame: 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: log CFU/g
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
log CFU/g
  GI Viability of Bacillus Spores Week 1 | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 1.2 (0.2)
  GI Viability of Bacillus Spores Week 5 | 1.1 (0.1) | 4.6 (0.1) | 5.6 (0.1) | 6.4 (0.1)
  GI Viability of Bacillus Spores Week 6 | 1.6 (0.1) | 1.3 (0.2) | 0.8 (0.1) | 2.1 (0.1)

3. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Cephalic
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Cephalic) Week 1 | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.04) | 0.2 (0.1)
  Daily Questionnaire (Cephalic) Week 2 | 0.2 (0.1) | 0.2 (0.1) | 0.1 (0.04) | 0.2 (0.1)
  Daily Questionnaire (Cephalic) Week 3 | 0.2 (0.1) | 0.2 (0.1) | 0.1 (0.04) | 0.3 (0.1)
  Daily Questionnaire (Cephalic) Week 4 | 0.4 (0.1) | 0.1 (0.03) | 0.2 (0.1) | 0.3 (0.1)
  Daily Questionnaire (Cephalic) Week 5 | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
  Daily Questionnaire (Cephalic) Week 6 | 0.2 (0.1) | 0.3 (0.1) | 0.2 (0.1) | 0.2 (0.1)

4. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Epidermal
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Epidermal) Week 1 | 0.1 (0.02) | 0.1 (0.1) | 0.01 (0.01) | 0.03 (0.01)
  Daily Questionnaire (Epidermal) Week 2 | 0.1 (0.04) | 0.02 (0.01) | 0.04 (0.02) | 0.04 (0.02)
  Daily Questionnaire (Epidermal) Week 3 | 0.04 (0.03) | 0.1 (0.1) | 0.1 (0.04) | 0.05 (0.03)
  Daily Questionnaire (Epidermal) Week 4 | 0.1 (0.04) | 0.02 (0.01) | 0.1 (0.1) | 0.04 (0.02)
  Daily Questionnaire (Epidermal) Week 5 | 0.1 (0.04) | 0.02 (0.01) | 0.02 (0.02) | 0.02 (0.02)
  Daily Questionnaire (Epidermal) Week 6 | 0.1 (0.04) | 0.02 (0.02) | 0.01 (0.01) | 0.02 (0.02)

5. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Ear, Nose, and Throat (ENT)
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (ENT) Week 1 | 0.2 (0.1) | 0.1 (0.4) | 0.1 (0.04) | 0.1 (0.04)
  Daily Questionnaire (ENT) Week 2 | 0.3 (0.2) | 0.4 (0.1) | 0.1 (0.03) | 0.1 (0.04)
  Daily Questionnaire (ENT) Week 3 | 0.3 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
  Daily Questionnaire (ENT) Week 4 | 0.4 (0.2) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
  Daily Questionnaire (ENT) Week 5 | 0.3 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
  Daily Questionnaire (ENT) Week 6 | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.1 (0.1)

6. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Behavioral
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Behavioral) Week 1 | 0.5 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.5 (0.1)
  Daily Questionnaire (Behavioral) Week 2 | 0.4 (0.1) | 0.2 (0.1) | 0.1 (0.1) | 0.6 (0.2)
  Daily Questionnaire (Behavioral) Week 3 | 0.4 (0.2) | 0.1 (0.1) | 0.1 (0.1) | 0.5 (0.1)
  Daily Questionnaire (Behavioral) Week 4 | 0.4 (0.2) | 0.1 (0.1) | 0.2 (0.01) | 0.5 (0.1)
  Daily Questionnaire (Behavioral) Week 5 | 0.6 (0.2) | 0.2 (0.1) | 0.1 (0.1) | 0.5 (0.2)
  Daily Questionnaire (Behavioral) Week 6 | 0.4 (0.1) | 0.3 (0.2) | 0.2 (0.1) | 0.5 (0.2)

7. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Emetic
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Emetic) Week 1 | 0.05 (0.04) | 0.003 (0.003) | 0.1 (0.1) | 0.1 (0.2)
  Daily Questionnaire (Emetic) Week 2 | 0.1 (0.1) | 0.1 (0.04) | 0.1 (0.04) | 0.03 (0.01)
  Daily Questionnaire (Emetic) Week 3 | 0.1 (0.04) | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  Daily Questionnaire (Emetic) Week 4 | 0.1 (0.1) | 0.02 (0.02) | 0.1 (0.1) | 0.1 (0.04)
  Daily Questionnaire (Emetic) Week 5 | 0.1 (0.1) | 0.1 (0.03) | 0.1 (0.1) | 0.03 (0.02)
  Daily Questionnaire (Emetic) Week 6 | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1) | 0.08 (0.04)

8. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Constipation
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Constipation) Week 1 | 0.2 (0.1) | 0.1 (0.1) | 0.4 (0.2) | 0.4 (0.2)
  Daily Questionnaire (Constipation) Week 2 | 0.1 (0.04) | 0.2 (0.1) | 0.3 (0.1) | 0.7 (0.3)
  Daily Questionnaire (Constipation) Week 3 | 0.3 (0.1) | 0.2 (0.01) | 0.3 (0.1) | 0.6 (0.2)
  Daily Questionnaire (Constipation) Week 4 | 0.3 (0.1) | 0.1 (0.1) | 0.6 (0.2) | 0.7 (0.3)
  Daily Questionnaire (Constipation) Week 5 | 0.2 (0.1) | 0.1 (0.1) | 0.5 (0.1) | 0.7 (0.2)
  Daily Questionnaire (Constipation) Week 6 | 0.3 (0.1) | 0.1 (0.03) | 0.5 (0.2) | 0.5 (0.2)

9. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Diarrhea
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Diarrhea) Week 1 | 0.2 (0.1) | 0.1 (0.04) | 0.2 (0.1) | 0.2 (0.1)
  Daily Questionnaire (Diarrhea) Week 2 | 0.2 (0.1) | 0.2 (0.03) | 0.2 (0.1) | 0.1 (0.03)
  Daily Questionnaire (Diarrhea) Week 3 | 0.2 (0.1) | 0.1 (0.1) | 0.3 (0.1) | 0.3 (0.1)
  Daily Questionnaire (Diarrhea) Week 4 | 0.2 (0.1) | 0.1 (0.1) | 0.4 (0.1) | 0.3 (0.1)
  Daily Questionnaire (Diarrhea) Week 5 | 0.4 (0.1) | 0.2 (0.1) | 0.3 (0.1) | 0.1 (0.1)
  Daily Questionnaire (Diarrhea) Week 6 | 0.3 (0.1) | 0.1 (0.04) | 0.2 (0.1) | 0.2 (0.1)

10. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Fatigue
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Fatigue) Week 1 | 1.1 (0.3) | 0.7 (0.2) | 0.7 (0.2) | 0.8 (0.2)
  Daily Questionnaire (Fatigue) Week 2 | 0.9 (0.3) | 0.6 (0.2) | 0.7 (0.2) | 0.9 (0.2)
  Daily Questionnaire (Fatigue) Week 3 | 0.9 (0.3) | 0.6 (0.2) | 0.7 (0.2) | 0.9 (0.2)
  Daily Questionnaire (Fatigue) Week 4 | 1.0 (0.3) | 0.4 (0.1) | 0.6 (0.2) | 0.9 (0.3)
  Daily Questionnaire (Fatigue) Week 5 | 0.8 (0.3) | 0.5 (0.1) | 0.6 (0.2) | 0.8 (0.2)
  Daily Questionnaire (Fatigue) Week 6 | 0.6 (0.3) | 0.5 (0.2) | 0.5 (0.2) | 0.7 (0.2)

11. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Satiety
Description: as for outcome 1
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Satiety) Week 1 | 0.8 (0.2) | 0.7 (0.2) | 0.9 (0.2) | 0.9 (0.2)
  Daily Questionnaire (Satiety) Week 2 | 0.7 (0.2) | 0.3 (0.1) | 0.8 (0.2) | 1.1 (0.3)
  Daily Questionnaire (Satiety) Week 3 | 0.9 (0.3) | 0.3 (0.1) | 0.8 (0.2) | 0.9 (0.2)
  Daily Questionnaire (Satiety) Week 4 | 0.9 (0.3) | 0.3 (0.1) | 0.8 (0.2) | 1.0 (0.3)
  Daily Questionnaire (Satiety) Week 5 | 0.9 (0.3) | 0.4 (0.1) | 0.9 (0.3) | 0.9 (0.3)
  Daily Questionnaire (Satiety) Week 6 | 0.8 (0.3) | 0.3 (0.1) | 0.9 (0.3) | 0.8 (0.3)

12. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Bowel Movement
Description: Daily Questionnaires consists of 24 symptom items evaluating general wellness. Participants filled out questionnaires nightly for the entire duration of the study (6 weeks). Daily scores were then averaged into weekly scores for each participant. Daily scores from weeks 2 - 5 were then averaged to arrive at a single value. Rating is scored from 0 (no symptoms) to 6 (very severe symptoms).
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  Daily Questionnaire (Bowel Mov.) Week 1 | 1.55 (0.2) | 1.5 (0.2) | 1.3 (0.1) | 1.5 (0.1)
  Daily Questionnaire (Bowel Mov.) Weeks 2-5 | 1.4 (0.1) | 1.5 (0.1) | 1.5 (0.1) | 1.5 (0.1)
  Daily Questionnaire (Bowel Mov.) Week 6 | 1.5 (0.2) | 1.4 (0.1) | 1.4 (0.1) | 1.6 (0.2)

13. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Wellness Questionnaires for Hours of Sleep
Description: Daily Questionnaires consists of 24 symptom items evaluating general wellness. Participants filled out questionnaires nightly for the entire duration of the study (6 weeks). Daily scores were then averaged into weekly scores for each participant. Participants recorded the number of hours they slept on the daily questionnaire.
Time Frame: Weekly for 6 weeks
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
Hours
  Daily Questionnaire (Hours of Sleep) Week 1 | 6.8 (0.2) | 6.6 (0.2) | 7.1 (0.1) | 6.6 (0.2)
  Daily Questionnaire (Hours of Sleep) Week 2 | 6.7 (0.1) | 6.8 (0.2) | 7.1 (0.2) | 6.9 (0.2)
  Daily Questionnaire (Hours of Sleep) Week 3 | 6.5 (0.2) | 6.8 (0.2) | 7.1 (0.2) | 6.7 (0.2)
  Daily Questionnaire (Hours of Sleep) Week 4 | 6.6 (0.2) | 7.0 (0.2) | 7.3 (0.2) | 6.8 (0.2)
  Daily Questionnaire (Hours of Sleep) Week 5 | 6.8 (0.2) | 7.0 (0.2) | 6.9 (0.2) | 6.9 (0.2)
  Daily Questionnaire (Hours of Sleep) Week 6 | 6.8 (0.2) | 7.0 (0.2) | 7.1 (0.1) | 6.7 (0.2)

14. Primary Outcome: Evaluation of the Effect of B. Subtilis R0179 on Gastrointestinal Symptoms Using Questionnaires
Description: Gastrointestinal Symptom Questionaires (GSRS) was administered during weeks 1, 5, and 6 of the study to evaluate gastrointestinal symptoms. The scale ranges from 1 (no discomfort at all) to 7 (very severe discomfort).
Time Frame: Weeks 1, 5, and 6
Population: Participants who completed all study requirements were included in the baseline analysis population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Number analyzed (Participants) | 20 | 21 | 20 | 20
units on a scale
  GSRS (Abdominal Pain) Week 1 | 1.6 (0.1) | 1.3 (0.1) | 1.4 (0.1) | 1.5 (0.2)
  GSRS (Abdominal Pain) Week 5 | 1.8 (0.1) | 1.5 (0.1) | 1.6 (0.1) | 1.6 (0.1)
  GSRS (Abdominal Pain) Week 6 | 1.7 (0.1) | 1.6 (0.2) | 1.6 (0.1) | 1.3 (0.1)
  GSRS (Reflux) Week 1 | 1.3 (0.1) | 1.3 (0.2) | 1.1 (0.1) | 1.1 (0.1)
  GSRS (Reflux) Week 5 | 1.3 (0.1) | 1.3 (0.2) | 1.1 (0.1) | 1.2 (0.1)
  GSRS (Reflux) Week 6 | 1.3 (0.1) | 1.3 (0.2) | 1.1 (0.1) | 1.2 (0.1)
  GSRS (Indigestion) Week 1 | 1.8 (0.1) | 1.4 (0.1) | 1.5 (0.01) | 1.7 (0.1)
  GSRS (Indigestion) Week 5 | 1.9 (0.2) | 1.6 (0.1) | 1.9 (0.1) | 1.6 (0.1)
  GSRS (Indigestion) Week 6 | 1.9 (0.1) | 1.3 (0.1) | 1.6 (0.1) | 1.7 (0.1)
  GSRS (Constipation) Week 1 | 1.5 (0.1) | 1.1 (0.1) | 1.4 (0.1) | 1.4 (0.1)
  GSRS (Constipation) Week 5 | 1.6 (0.1) | 1.2 (0.1) | 1.6 (0.2) | 1.8 (0.2)
  GSRS (Constipation) Week 6 | 1.5 (0.1) | 1.2 (0.1) | 1.6 (0.2) | 1.7 (0.2)
  GSRS (Diarrhea) Week 1 | 1.3 (0.1) | 1.2 (0.1) | 1.3 (0.2) | 1.4 (0.1)
  GSRS (Diarrhea) Week 5 | 1.7 (0.2) | 1.2 (0.1) | 1.6 (0.2) | 1.5 (0.1)
  GSRS (Diarrhea) Week 6 | 1.8 (0.2) | 1.3 (0.1) | 1.4 (0.2) | 1.3 (0.1)

ADVERSE EVENTS:
Time Frame: Data monitoring adverse events was collected over the study period.
Arm/Group | Placebo | B. Subtilis R0179 (0.1 Billion CFU) | B. Subtilis R0179 (1 Billion CFU) | B. Subtilis R0179 (10 Billion CFU)
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/22 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | B. Subtilis R0179 (0.1 Billion CFU) (N=21) | B. Subtilis R0179 (1 Billion CFU) (N=22) | B. Subtilis R0179 (10 Billion CFU) (N=20)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One participant reported a serious adverse event of hospitalization with an admitting diagnosis of hypotension, but did not discontinue probiotic consumption and completed the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | B. Subtilis R0179 (0.1 Billion CFU) (N=21) | B. Subtilis R0179 (1 Billion CFU) (N=22) | B. Subtilis R0179 (10 Billion CFU) (N=20)
Diarrheal Symptoms (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One participant in the 0.1 billion CFU treatment group experienced diarrheal symptoms and completed the study, this event did not occur in any other participants and did not persist.
Itchiness and Redness Symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — A participant in the 10 billion CFU treatment group experienced itchiness/redness symptoms that were sporadic and persisted for several days. The participant voluntarily withdrew from the study, these symptoms did not occur in any other participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No